CLINICAL TRIAL: NCT07285070
Title: A Phase 2, Randomized, Double-Masked, Controlled, Proof-of-Concept Study to Evaluate the Safety and Biological Activity of a Water-free Tacrolimus Ophthalmic Solution (NOV05) for the Treatment of Non-Infectious Anterior Uveitis
Brief Title: Tacrolimus Ophthalmic Solution for the Treatment of Non-infectious Anterior Uveitis
Acronym: EYETAC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NOV05-001
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-infectious Anterior Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tacrolimus ophthalmic solution (high dose) (Active Comparator)
  Interventions: Drug: Tacrolimus ophthalmic solution
- Tacrolimus ophthalmic solution (low dose) (Active Comparator)
  Interventions: Drug: Tacrolimus ophthalmic solution

INTERVENTIONS:
Drug: Tacrolimus ophthalmic solution — high and low dose treatment will be compared over 6 weeks treatment

SUMMARY:
The primary objective of the study is to investigate the safety and tolerability of NOV05 eye drops at two concentrations QID in patients with active non-infectious anterior uveitis.

DETAILED DESCRIPTION:
This first in-human, phase 2 proof of concept study aims to show that the formulation at two concentrations is safe and well tolerated over a period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years of age;
* Provide written informed consent;
* Be diagnosed with active non-infectious anterior uveitis requiring initiation or increase of topical steroids administration for the management of ocular inflammation;
* Have an onset of symptoms within 4 weeks;

Exclusion Criteria:

* Have severe/serious ocular pathology in the study eye which may preclude study completion or interferes with trial assessment, in the judgement of the clinical Investigator;
* Have a history of or a current ocular or periocular malignancy;
* Have active intermediate or posterior uveitis in the study eye or another documented posterior segment inflammation;
* A confirmed or highly suspicious infectious uveitis eg, CMV, Herpes simplex, Herpes zoster, syphilis, tuberculosis, lyme disease;
* Have a known allergy or sensitivity to the IMP tacrolimus or semifluorinated alkanes (SFA);
* Be a woman who is pregnant, nursing, or planning a pregnancy;
* Have a condition or be in a situation (e.g. language barrier, non-cooperative, history of substance abuse) which the Investigator considers that it may put the patient at significant risk, may confound the trial results, or may significantly interfere with the patient's participation in the trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 8 weeks
  ocular and non-ocular adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, PhD, Study Director — Novaliq GmbH

IPD SHARING:
Plan to Share IPD: No